CLINICAL TRIAL: NCT05671991
Title: Effect of Empagliflozin on Peritoneal and Kidney Function in End Stage Renal Disease
Acronym: EMPA-PD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000031605
Record Dates: First submitted 2022-12-14; First posted 2023-01-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Peritoneal dialysis
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, acute crossover study of empagliflozin in 30 chronic PD patients, with an 8 week "pre post" open label extension in all 30 patients where they will receive empagliflozin daily.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin or Placebo in Acute (Experimental): Acute phase: Participants will receive 25 mg empagliflozin once on Day 0 or Day 7. Participants receive empaglifozin or placebo on Day 0. On Day 7, they will be crossed over to the alternate treatment.
  Interventions: Drug: Empagliflozin 25 mg vs Placebo
- Empagliflozin in Chronic (Active Comparator): Chronic phase: On day 8, all participants will receive 10 mg empagliflozin 10 mg x 8 weeks
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 25 mg vs Placebo — Acute Study- Empagliflozin 25 mg vs Placebo on D1 then alternate therapy on D7
  Arms: Empagliflozin or Placebo in Acute
Drug: Empagliflozin 10 MG — Chronic Study- Empagliflozin 10 mg for 8 weeks
  Arms: Empagliflozin in Chronic

SUMMARY:
The main purpose of the study is to determine if empagliflozin can reduce peritoneal glucose absorption in patients with end stage renal diease (ESRD) on peritoneal dialysis.

This is a randomized, placebo controlled, acute crossover study of empagliflozin in an anticipated 30 chronic PD patients, with an 8 week "pre post" open label extension in all 30 patients where they will receive empagliflozin daily.

DETAILED DESCRIPTION:
Participants will undergo three study visits, and up to 4 safety visits, over 9 weeks.

At 7 AM in the first study visit, the participants will have taken 25mg empagliflozin once or matching placebo, thus producing peak plasma levels by 10 AM. One week later the participant will return for the crossed over to the alternate study drug.

At the conclusion of the 2nd study visit, all participants will be provided with empagliflozin 10mg tabs to be taken daily for 56 days (8 weeks). At each study visit and safety visit, participants will undergo a PET test.

ELIGIBILITY:
Inclusion Criteria

1. Patients actively undergoing PD with a reliably functioning PD catheter
2. Stable peritoneal dialysis prescription
3. PD vintage > 3 months
4. Age >18 years of age

Exclusion Criteria:

1. History of type 1 diabetes, diabetic ketoacidosis, "brittle" diabetes or frequent hypoglycemia or severe hypoglycemic episodes requiring emergent intervention (ER visit or EMS response, glucagon administration or forced oral carbs) in the last 6 months
2. Use of an SGLT2 inhibitor within the prior 30 days
3. 1 or more episodes of peritonitis in the previous 6 months or active infection of the peritoneal dialysis catheter
4. Anemia with hemoglobin <8g/dL
5. Inability to give written informed consent or follow study protocol
6. Contraindication to receiving loop diuretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Glucose absorption with empagliflozin vs. placebo | Day 0 to Day 63
  Total glucose absorption in grams with empagliflozin vs. placebo

SECONDARY OUTCOMES:
Ultrafiltration volume with empagliflozin vs. placebo- acute study | at 4 hours
  Ultrafiltration volume (in liters) at 4 hours with empagliflozin vs. placebo.
Change in plasma glucose levels with empagliflozin vs. placebo- acute study | Day 0 to Day 63
  Change in plasma glucose levels during PD dwell with empagliflozin vs. placebo- acute study
Increase in natriuresis with empagliflozin vs. placebo-acute study | Day 0 to Day 63
  Natriuresis determined by FENa
Change in peritoneal fluid inflammatory markers | Day 0 to Day 63
  Change in levels of IL-6 and CA-125 (in pg)
Change in PET test parameters | Day 0 to Day 63
  Change in peritoneal equilibration test parameters, measurement of solute transport across the peritoneal membrane (standard test carried out in PD patients to assess solute trasnport across membrane)
Change in total body water and extracellular water | Day 0 to Day 63
  Change in total body water and extracellular water, using heaving water (D20)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States